CLINICAL TRIAL: NCT03955068
Title: Pilot Study of a Strict Classic Ketogenic Diet as a Therapy for Recurrent or Progressive and Refractory Brain Tumors in Children
Brief Title: Strict Classic Ketogenic Diet as a Therapy for Recurrent or Progressive and Refractory Brain Tumors in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding for this study.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Bowers, Professor of Pediatrics Hematology/Oncology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-0853
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Brain Tumor, Childhood; Ketogenic Diet
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strict Classic Ketogenic Diet Arm (Other): The classic ketogenic diet is individually calculated for each patient based on age, weight, and nutritional needs. The diet is typically administered from a 2:1 to 4:1 ratio; this means 2 to 4 parts of fat to 1 part of both protein (calculated based on RDA and whatever remaining portion of carbohydrates. The basis of calculations is first on the amount of required protein needed to meet RDA to insure adequate growth. Fine tuning of ketogenic diet therapy is based on serum beta-hydroxybutyrate levels (target levels of 3.5-6.5 mmol/L), tolerance of the diet, and response to treatment.
  Interventions: Other: Strict Classic Ketogenic Diet

INTERVENTIONS:
Other: Strict Classic Ketogenic Diet — Diet is administered from a 2:1 to 4:1 ratio; this means 2 to 4 parts of fat to 1 part of both protein (calculated based on RDA and whatever remaining portion of carbohydrates.

SUMMARY:
This is a pilot study to test the feasibility of implementing a strict classic ketogenic diet among a population of children with recurrent or progressive and refractory brain tumors. Eligible participants will be admitted to the neurosciences floor for 5 days to begin the ketogenic diet either orally, by gastrostomy tube or via nasogastric tube. During the inpatient stay, they will be extensively educated on the diet restrictions and rules. Participants will then continue on the diet at home returning about 17 times over the next 12 months. Daily logs will be kept tracking diet changes, bowel movements and urine ketones. Blood will be collected during the inpatient stay and at all visits for both standard clinical care and research testing.

DETAILED DESCRIPTION:
Primary Objective is to determine the feasibility (safety and tolerability) of a strict classic ketogenic diet among a population of children with recurrent or progressive and refractory brain tumors.

Secondary Objectives are: (1) to determine the objective response rate (complete response + partial response) to a strict classic ketogenic diet among children with recurrent or progressive and refractory brain tumor; (2) to estimate the time interval to tumor progression (Progression-Free Survival), time to treatment failure (Event-Free Survival), and time to death (Overall Survival) after initiation of a strict classic ketogenic diet among a group of pediatric patients with recurrent or progressive and refractory brain tumors; and (3) to describe and characterize tolerability and toxicities from a strict classic ketogenic diet among children with recurrent or progressive and refractory brain tumors.

Exploratory Objective: Identify biomarker correlates, including MR spectroscopy and metabolites of tumor response to a strict classic ketogenic diet.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be < 21 years of age inclusive at the time of enrollment on this protocol.
* Histologic Diagnosis: Histologically proven, primary brain tumor that is recurrent or progressive and refractory (nonresponsive) to standard, accepted therapy. A histopathologic diagnosis from either the initial presentation or at the time of recurrence is required for all subjects, except for diffuse intrinsic pontine glioma (DIPG).
* Measurable Disease: Patients must have radiographically documented measurable tumor as assessed by RANO or RAPNO criteria.
* Cranial and Spinal MRI: To document the degree of residual tumor, all patients must have an MRI of the brain with and without gadolinium performed within 2 weeks prior to study enrollment. For patients who undergo a tumor debulking surgery at the time of recurrence/progression, the following must be obtained:
* Cranial pre-operative MRI scan with and without contrast.
* Cranial post-operative MRI scan with and without contrast within 28 days following surgery. If possible, post-operative MRI should be performed within 48 hours of surgery, prior to the onset of edema or post-operative surgical enhancement, which can make measurements of residual tumor difficult.
* Performance Level: Patients must have a performance status of > 50. Use Karnofsky score for patients > 16 years of age and Lansky score for patients ≤ 16 years of age.
* Life Expectancy: Patients must have a life expectancy of > 8 weeks.
* Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, biologic therapy, or radiotherapy prior to entering this study
* Growth factor(s): Must not have received within 1 week prior to entry onto this study.
* Other anti-cancer or experimental agents or therapies are not permitted. Homeopathic medicines are not permitted. Multivitamins are permitted.
* Organ Function Requirements: Adequate bone marrow, renal, liver, pulmonary, and central nervous system function
* All patients and/or their parents or legal guardians must sign a written informed consent.
* In the investigator's opinion, patients must have the ability to adhere to or tolerate the dietary protocol.
* Patients must be able to eat by mouth or must be willing to have a nasogastric tube (NGT) if gastrostomy tube is not already present.

Exclusion Criteria:

* Pregnancy
* Pregnant or breastfeeding. Female patients of childbearing potential must have negative pregnancy test result within the previous 14 days..
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation.
* Other Exclusionary Criteria: Disorder of B-oxidation, as measured by plasma aceyl-carnitine, Uncontrolled infection, History of nephrolithiasis, Diagnosis of diabetes mellitus that is being treated by medication.
* The following medications are excluded: Steroids: Therapeutic systemic doses of steroids must be stopped greater than 2 weeks prior to admission to the hospital to start the diet. A steroid washout of 1 week is acceptable for patients with DIPG. Concomitant chemotherapy drugs and homeopathic drugs are not permitted.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility (safety and tolerability) of the ketogenic diet | 28 days
  Defined by the enrolled subject completing 28 days of ketogenic diet therapy without grade 3 - 5 adverse events. These will be assessed via NCI's CTCAE v5.0 toxicity criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bowers, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States